

# High Intensity Functional Training in the Rehabilitation of Cancer Survivors

### Study protocol of a pragmatic clinical trial

Andreas Lund Hessner, PT, MSc

Henning Langberg, Professor

Jette Vibe-Petersen, MD

Karen Trier, PT, Msc

Maja S. Sommer, PT, PhD

Rikke Daugaard, PT, Msc

Rasmus Tolstrup Larsen, PT, MSc

Date: June 26, 2019

Clinical trials ID: 514-0306/19-3000

### Title page

| 1 | Title |
|---|---|
| 2 | High Intensity Functional Training in the rehabilitation of cancer survivors: Study protocol of a |
| 3 | pragmatic clinical trial |
| 4 | |
| 5 | Corresponding and first author: Andreas L. Hessner <sup>1</sup> , PT, MSc. (hessnerfysioterapi@gmail.com) |
| 6 | Henning Langberg <sup>1</sup> |
| 7 | Jette Vibe-Petersen <sup>2</sup> |
| 8 | Karen Trier <sup>2</sup> |
| 9 | Maja S. Sommer <sup>2</sup> |
| 10 | Rikke Daugaard <sup>2</sup> |
| 11 | Rasmus T. Larsen <sup>1</sup> , PT, MSc. (rala@sund.ku.dk) |
| 12 | |
| 13 | Affiliation |
| 14 | <sup>1</sup> CopenRehab, Section of Social Medicine, Dept. of Public Health, |
| 15 | University of Copenhagen, Henrik Pontoppidansvej 6, 1., 2200 Copenhagen N. |
| 16 | <sup>2</sup> Centre for Cancer and Health Copenhagen, Nørre Allé 45, 2200 Copenhagen N. |
| 17 | |
| 18 | Text word count: 2922 |
| 19 | Keywords: Crossfit, High Intensity Functional Training, Cancer, Cancer survivors |
| 20 | |
| 21 | |
| 22 | |
| 23 | |
| 24 | |
| 25 | |
| 26 | |
| 27 | |
| <ul><li>28</li><li>29</li></ul> | |
| 30 | |
| 31 | |

| 32 | Table of contents |
|---|---|
| 33 | TITLE |
| 34 | BACKGROUND AND RATIONALE |
| 35 | OBJECTIVE4 |
| 36<br>37<br>38<br>39<br>40<br>41<br>42<br>43 | METHODS: PARTICIPANTS INTERVENTIONS AND OUTCOMES5DESIGN AND STUDY SETTING5ELIGIBILITY CRITERIA5INTERVENTION6PATIENT-REPORTED OUTCOMES7Primary outcomes7Secondary outcomes8RECRUITMENT9 |
| 44 | METHODS: DATA COLLECTION, MANAGEMENT AND ANALYSIS |
| 45<br>46 | Data collection methods |
| 47 | STATISTICAL METHODS |
| 48<br>49<br>50<br>51 | ETHICS AND DISSEMINATION |
| 52 | AUTHORS CONTRIBUTIONS |
| 53 | REFERENCES |
| <ul><li>54</li><li>55</li><li>56</li><li>57</li><li>58</li></ul> | APPENDIX 1 |
| 59 | Background and rationale |
| 60 | Cancer survivors experience a variety of ongoing physical and psychological symptoms associated |
| 61 | with both disease and treatment (1,2). Additionally, cancer survivors have an increased risk of |
| 62 | serious chronic health sequelae and comorbid conditions such as cardiovascular disease and |
| 63 | diabetes (2). These poor health outcomes among cancer survivors have led to greater emphasis on |
| 64 | interventions to enhance health outcomes such as health-related quality of life (HRQoL) and |
| 65 | cancer-related fatigue (CRF) (3). |
| 66 | Aerobic training as well as resistance training are both exercise interventions associated with a |
| 67 | |
| | number of health benefits in survivors of a variety of cancers (4–7). Thus, clinical guidelines |

69 rehabilitation of cancer survivors during and after active cancer treatment (1,8,9). 70 Furthermore, aerobic training and resistance training performed at high intensity has been reported 71 as a feasible and safe intervention for patients with various different cancer diagnosis and in 72 different stages of cancer. It can provide objective physiological benefits as well as improve 73 HRQoL, CRF and depression among cancer survivors (4,5,7,10–12). 74 High Intensity Functional Training (HIFT) has been defined as a style of training that incorporates 75 functional, multimodal movements, performed at relatively high intensity, and designed to improve 76 parameters of general physical fitness and performance (13). In recent years HIFT has gained 77 increasing attention in the fitness industry and in research (14), especially due to the increased 78 popularity of the HIFT program CrossFit© (13). Recently trials, using HIFT protocols, have 79 reported benefits in healthy adults including physiological improvements such as increased oxygen 80 consumption, improved body composition and bone health (15,16). 81 One identified study by Heinrich et al examined the effectiveness and feasibility of 5 weeks of 82 HIFT among cancer survivors with a variety of cancer diagnoses. The study included 8 participants 83 and reported that the intervention was well-received, feasible and associated with a significant 84 improvement in emotional functioning and body composition. 85 HIFT is viewed as a promising type of training (13,17), that has shown numerous physiological 86 benefits (15,16,18) and has shown preliminary effectiveness and feasibility among cancer survivors 87 (17).88 Furthermore, several reports and clinical guidelines recommend the prescription of exercise 89 programs that are enjoyable and facilitates social interactions, motivation and continued 90 participation to reduce risk of the development of comorbid conditions and late-appearing effects 91 of cancer and its treatment (1,8,19). HIFT has been reported to be associated with higher levels of enjoyment than more traditional resistance training, and to facilitate adherence, continued 92 93 participation and sense of community among healthy participants (18,20). 94

### **Objective**

95

- The primary objective of this pragmatic clinical trial is to test the feasibility of the intervention in a
- 97 real world setting and secondary, to describe whether the HRQoL of the participants changes from
- baseline to end-point and follow up time points. Furthermore, we will investigate the association
- between the leisure-time HIFT and the HRQoL.

| 100 | |
|---|---|
| 101 | Methods: Participants interventions and outcomes |
| 102 | This study protocol is reported according to the Guidelines for Inclusion of Patient-Reported |
| 103<br>104 | Outcomes in Clinical Trial Protocols (SPIRIT-PRO) Extension. |
| 105 | Design and study setting |
| 106 | This study is a single group clinical trial. A pragmatic design will be applied for this study to |
| 107 | increase transferability, generalizability and the external validity of the results into clinical practise. |
| 108 | Thus, the clinical setting for the intervention will be at the municipality rehabilitation centre, Centre |
| 109 | for Cancer and Health Copenhagen (CCHC), in the capitol region of Denmark. |
| 110 | The exercise intervention will be implemented as a part of regular practice at the centre and will be |
| 111 | supervised by CCHC's physiotherapists. Two co-authors of this protocol (MS and RD) are |
| 112 | employed as physiotherapists at CCHC. They have contributed in designing this study to fit the |
| 113 | clinical reality and the specific patient group at CCHC. This is another way increasing the external |
| 114 | validity of the results of this study, and to 'bridge the gap' between research and clinical practise. |
| 115 | This implementation of community-based clinicians in physiotherapy research has previously been |
| 116 | recommended in the literature (21,22). |
| 117 | |
| 118 | Eligibility criteria |
| 119 | Due to the pragmatic design of this study, only few inclusion- and exclusion criteria will be applied |
| 120 | Patients will be considered eligible for inclusion when they; 1) are at least 18 years old, 2) are |
| 121 | referred to the centre for cancer rehabilitation from any hospital or private practising general |
| 122 | practitioner in the Capital Region in Denmark, 3) Choosing to participate in group based high |
| 123 | intensity functional training that is offered at CCHC as part of their physical rehabilitation. |
| 124 | Eligibility for participation in this study will be regardless of cancer treatment and the stage of the |
| 125 | cancer. Thus, both patients undergoing active cancer treatment, patient who have completed active |
| 126 | treatment as well as chronic cancer survivors will be considered eligible_for participation in this |
| 127 | study. |
| 128 | The following exclusion criteria will be applied for this study: 1) Not able to reply to the |
| 129 | questionnaire due to mental impairment, 2) Patients who are not able to read and understand |

160

130 Danish, 3) Patients who does not have an e-mail address because of the application of online-based 131 questionnaires. 132 Intervention 133 The exercise intervention for this study will be HIFT, as defined by Feito et al and described in the 134 introduction of this study protocol (13). The program design and template will be based on the 135 principles of the HIFT program called CrossFit®. CrossFit is described as a strength and 136 conditioning program that focuses on "constantly varying functional movements, performed at a 137 relatively high intensity" (23). CrossFit training includes a variety of elements from gymnastics 138 (e.g., floor, bar and ring exercises), weightlifting exercises (e.g., squats, cleans, snatches and presses 139 with a barbell, dumbbell or kettlebell), and cardiovascular activities (e.g., running or rowing) (24). 140 141 142 All group training sessions will take place in a clinical setting at CCHC. 143 The full exercise protocol template is designed as a 38-week HIFT program, as the inclusion of 144 participants will be consecutive. All participants will complete 16 weeks of twice weekly groupbased HIFT sessions, under the supervision of two physiotherapists, specifically trained to deliver 145 146 the HIFT program. Given the consecutive nature of this inclusion process, the participants will initiate the group-based training at different dates between august 5<sup>th</sup> 2019 and January 5<sup>th</sup> 2019 (see 147 148 figure 2 for process of HIFT program implementation and figure 3 for timeline of the study period with important dates). 149 150 151 Each training session will last for one hour and 15 minutes and will include a general warmup, a 152 strength-focused section including 1-3 exercises and a aerobic-focused workout. 153 The exercise program is not developed to include a general progression in terms of resistance, 154 intensity or volume over the cause of 38 weeks. An exercise compendium will be developed to meet 155 one of the key principles of CrossFit, that is scalability (25). The compendium will include 156 movement standards as well as progressions and regressions of all included exercises. This is to 157 assist the supervising physiotherapists in choosing the relevant level of intensity and exercise difficulty for each participant, and to allow for individual progression over the cause of the 16-week 158 159 exercise intervention period for each participant.

| 161 | Patient-reported outcomes |
|---|---|
| 162 | EORTC: |
| 163 | EORTC QLQ-C-30 includes five functional domains (physical, role, cognitive, emotional and |
| 164 | social, where higher scores represent greater function or quality of life) and three symptom scales |
| 165 | (fatigue, pain and nausea). Functional and symptom scales range from 0 to 100. Higher values on |
| 166 | functional scales equal a higher level of functioning. Higher values on symptom scales equal higher |
| 167 | symptom burden. EORTC QLQ-C-30 is chosen for it's established reliability and validity with |
| 168 | specific emphasis on use in cancer populations (26, 27). |
| 169 | GLTEQ: |
| 170 | Leisure time physical activity (LTPA) will be assessed using an original Danish translation of the |
| 171 | Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ) .The GSLTPAQ is |
| 172 | frequently used in oncology research to assess LTPA. |
| 173 | The GSLTPAQ is a 4-item self-administered questionnaire. The first three questions ask for |
| 174 | information on the number of times the respondant engages in mild, moderate and strenuous LTPA |
| 175 | bouts of at least 15 min duration in a typical week. A score is then calculated for total leisure time |
| 176 | based on the numerical values attributed to each of the three categories (9 for strenuous, 5 for |
| 177 | moderate and 3 for light) multiplied by the frequency of the activity. The scores derived from this |
| 178 | method is called a Leisure Score Index (LSI). In addition, scores obtained from moderate and |
| 179 | strenuous physical activity can be used to classify respondents into active and insufficiently active |
| 180 | categories. |
| 181 | A recently published systematic review by Amireault et al, supports the use of the GSLTPAQ in |
| 182 | oncology research and the interpretation of the LSI for assessing relative change in PA among |
| 183 | cancer survivors. |
| 184 | |
| 185 | Primary outcomes |
| 186 | HRQoL will be evaluated using the Global Health Status/Quality of Life item from the EORTC |
| 187 | QLQ-C-30 questionnaire. The item ranges from 0 to 100, and higher values equal higher HRQoL. |
| 188 | Time frame: for each participant at baseline + end point at 16 weeks + follow up at 3 month and 12 |
| 189 | months) |

| 190 | |
|---|---|
| 191 | |
| 192 | Secondary outcomes |
| 193 | The secondary outcomes include functional scales (physical, role, emotional, cognitive, and social) |
| 194 | and symptom scales (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, |
| 195 | constipation, diarrhea, and financial difficulties) from the EORTC QLQ-C30 questionnaire). |
| 196 | In addition to the EORTC QLQ-C30 scales, leisure-time exercise will be included as a secondary |
| 197 | outcome and will be assessed using the GSLTPAQ, including the frequency and duration of mild, |
| 198 | moderate and strenuous exercise. |
| 199 | [Time frame for each participant: Baseline + end point at 16 weeks + follow up at 3 months and 12 |
| 200 | months] |
| 201 | Continued participation in any high intensity functional training (post-intervention HIFT) will be |
| 202 | assessed using a single-item modified version of the (GSLTPAQ) asking participants: During a |
| 203 | typical 7-Day period (a week), how many times on the average do you do High Intensity Functional |
| 204 | Training (I.E. CrossFit) for more than 15 minutes during your free time. The participant responds |
| 205 | by typing how many times per week, starting from zero. |
| 206 | [Time frame: for each participant at follow up at 3 month and 12 months] |
| 207 | |
| 208 | |
| 209 | Participation timeline |
| 210 | The inclusion of participants will be consecutive as patients are referred to CCHC for physical |
| 211 | cancer rehabilitation from various hospitals in the Capital Region in Denmark (see figure 1 for |
| 212 | participation flow of each participant). |
| 213 | Self-reported baseline data will be collected using online questionnaires sent out to patients via |
| 214 | email within four days prior to beginning the supervised HIFT intervention. After completing the 16 |
| 215 | weeks of high intensity functional training the patient will receive an end point questionnaire. |
| 216 | Three months following completing the exercise intervention, participants will be contacted via |
| 217 | email to complete a follow-up questionnaire also including questions regarding continued |
| 218 | participation in HIFT. All participants will receive an identical follow-up questionnaire 12 month |

| 219 | after completing the intervention. |
|---|---|
| 220 | |
| 221 | Sample size |
| 222 | Due to the exploratory nature of this study, no power calculation will be conducted. As the |
| 223 | inclusion of participants will be consecutive, the anticipated number of included participants will be |
| 224 | estimated based on the average monthly number of patients that begins the group based training |
| 225 | during clinical practise at the centre. The average number of patients who is referred to the |
| 226 | rehabilitation centre and who begins the HIFT training every month is 6 and thus, it is expected that |
| 227 | a total of approximately 30 participants will be included in this study during a 22-week consecutive |
| 228 | inclusion period that runs from august 5 <sup>th</sup> 2019 to January 5 <sup>th</sup> . All participants will be asked to |
| 229 | complete both baseline-, end point- and three-month follow-up assessment. |
| 230 | |
| 231 | Recruitment |
| 232 | Due to the pragmatic design there will be no recruitment though advertisement. Recruitment will |
| 233 | take place by asking eligible patients referred to CCHC, if they would like to participate in the |
| 234 | study. This recruitment will take place during an initial rehabilitation planning session with a |
| 235 | physiotherapist two days prior to the first HIFT session. Patients will be made aware that they have |
| 236 | two days to consider participating in the study (written participant information can be found in |
| 237 | appendix 1). |
| 238 | |
| 239 | Methods: Data collection, management and analysis |
| 240 | Data collection methods |
| 1<br>241 | Plan for assessment and collection of outcomes |
| 242 | All primary and secondary outcomes are participant-reported and will be administered through the |
| 243 | online survey tool: SurveyXact. All included participants will receive an email with an electronic |
| 244 | SurveyXact_invitation to the baseline questionnaire the same days as providing written consent to |
| 1<br>245 | participate in the study. On the day of the final HIFT session (week 16), the participants will receive |
| 246 | a similar SurveyXact_invitation with the end-point questionnaire. The three and 12-month follow up |
| 1<br>247 | assessments will be administered in identical ways to the end-point assessment. |

| 248 | |
|---|---|
| 249 | Patient characteristics |
| 250 | Demographic variables will be included in the baseline questionnaire. These will include self- |
| 251 | reported information about: sex, body mass index, educational level, employment, smoking status |
| 252 | and physical activity level, and will be collected together with information on cancer type, time |
| 253 | since cancer diagnosis, time since active treatment and cancer treatment type. |
| 254 | |
| 255 | Registration of adverse events, plans to promote participant retention and complete follow |
| 256 | up: |
| 257 | Adverse events and reasons for drop out from discontinued participant will be collected by |
| 258 | practising physiotherapists at CCHC. |
| 259 | To minimize non-response and loss to follow-up participants will receive a reminder by email 4 and |
| 260 | 14 days after receiving the email with end-point and follow-up questionnaire if they haven't |
| 261 | provided their responses. |
| 262 | |
| 263 | Data management |
| 264 | All outcomes will be handled and stored electronically on a secure server for personal data, located |
| 265 | at the University of Copenhagen. |
| 266 | No personal data will be exported from SurveyXact without pseudonymization. Complete |
| 267 | anonymization of all data will be done after the last follow up period. Data protection agency |
| 268 | approval Reference number: 514-0306/19-3000 |
| 269 | |
| 270 | Statistical methods |
| 271 | Descriptive statistics will be used to summarize patient characteristics including age, sex, cancer |
| 272 | diagnosis and type of treatment. Furthermore, leisure-time HIFT exercise and HRQoL at baseline |
| 273 | will be summarized using the GSLTPAQ LSI score and the EORTC QLQ-C30 GH score |
| 274 | respectively. Quantile Quantile plots and histograms will be used to evaluate distribution of |
| 275 | standardized residuals. Continous data with normally distributed standardized residuals will be |
| 276 | summarized using parametric statistics. Continous data with without normally distributed |
| 277 | standardized residuals will be summarized as ordinal data, using non-parametric statistics. |
| 278 | Categorical data will be summarized using frequencies and % of total. |

| 279 | The EORTC QLQ outcomes will be conducted according to the EORTC QLQ-C30 scoring manual |
|---|---|
| 280 | (ref fayes 2001). Numerical data for each outcome with normal distributed standardized residuals, |
| 281 | will be analysed from baseline to end-point with parametric statistics (paired t-test with equal |
| 282 | variance). Single-Factor Repeated Measures Design will be conducted with a repeated measures |
| 283 | one-way analysis of variance with four within subject time levels: baseline, end-point, three month |
| 284 | follow up, and 12-month follow up. Summary statistics will include mean and confidence intervals |
| 285 | for each outcome. |
| 286 | Numerical data for each outcome, without normal distributed standardized residuals, or ordinal data |
| 287 | will be analyzed from baseline to end-point with non-parametric statistics (Wilcoxon signed-ranks |
| 288 | test). Single-Factor Repeated Measures Design will be conducted with a Friedman two-way |
| 289 | analysis of variance by ranks with four within subject time levels: baseline, end-point, three months |
| 290 | follow up, and 12-month follow up. Summary statistics will include medians and interquartile |
| 291 | ranges for each outcome, and visualizations will include bar charts with confidence intervals. |
| 292 | The association between leisure-time HIFT exercise and HRQoL will be analyzed on each time |
| 293 | point with a linear regression model. To test whether the associations varies, the coefficients from |
| 294 | the linear regression analyses will be compared. |
| 295 | Stata 15.1 (StataCorp, College Station, TX, USA) will be used for all statistical analyses and |
| 296 | illustrations and an alpha level of 0.05 or less will be considered statistically significant. |
| 297 | |
| 298 | Ethics and dissemination |
| 299 | The study will be performed according to the Declaration of Helsinki. |
| 300 | The Regional Scientific Ethics Committee of Capitol Region in Denmark has reviewed the outline |
| 301 | of this study. The committee waived the need for ethical approval as the intervention in the study is |
| 302 | a part of the regular practice at the CCHC. Thus, the committee proclaimed that the study include |
| 303 | "no or minimal health intervention". Such studies can be implemented without permission from th |
| 304 | Ethics Committee according to Danish legislation (Committee Act § 2). |
| 305 | All included participants will provide written informed consent to participate in this study. |
| 306 | The study findings will be disseminated in peer reviewed journals and will be presented at national |
| 307 | conferences |

| 308 | |
|---|---|
| 309 | |
| 310 | Locations |
| 311 | Center for Kræft og Sundhed København, Capital Region, Denmark, 2200 Copenhagen N. |
| 312 | |
| 313 | Collaborators |
| 314 | Section of Social Medicine, Dept. of Public Health, Faculty of Health. University of Copenhagen. |
| 315 | Gothersgade 160, 3. sal |
| 316 | 1123 København K |
| 317 | |
| 318 | Principal investigator |
| 319 | Andreas Lund Hessner |
| 320 | |
| 321 | |
| 322 | Authors contributions |
| 323 | ALH (principle investigator. ALH is the study coordinator and is responsible for, data collection, developing the |
| 324 | exercise intervention program and drafting of the manuscript. ALH and RT are responsible for data analysis. All |
| 325 | authors contributed to the design of the study. All authors will edit and approve the final manuscript. |
| 326 | |
| 327 | Acknowledgements |
| <ul><li>328</li><li>329</li></ul> | No funds are present at current stage. |
| 330 | Abbreviations (In chronological order) |
| 331 | CS – Cancer Survivors |
| 332 | HRQoL – Health-related Quality of Life |
| 333 | CRF – Cancer-Related Fatigue |
| 334 | HIFT - High Intensity Functional Training |
| 335 | CKSK – Center for Kræft og Sundhed København (Center for Cancer and Health Copenhagen) |
| 336 | WOD – Workout of the Day |
| 337 | EORTC QLQ-C30 - European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 |
| 338 | GLTEQ – Godin Leisure-time Exercise Questionnaire |
| 339 | |
| 340 | Declarations of interests |
| 341 | ALH and RTL are both part time employees at the CrossFit affiliate CrossFit Copenhagen Aps. CrossFit Copenhagen |
| 342 | has supplied some additional exercise equipment for the intervention and offered the five supervising physiotherapists |
| 343 | from CCHC spots on their Trainers Course in order to develop and improve the physiotherapists HIFT-specific |

- instruction skills. ALH and RTL have not received any funds neither CrossFit Copenhagen or CCHC, nor will they
- during the conduction of this study. The study is not a part of ALH and RTL's occupation at CrossFit Copenhagen.

346

347

#### References

- 348 1. Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvão DA, Pinto
- 349 BM, et al. American College of Sports Medicine roundtable on exercise guidelines for cancer
- 350 survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409–26.
- 2. Pachman DR, Barton DL, Swetz KM, Loprinzi CL. Troublesome symptoms in cancer
- survivors: fatigue, insomnia, neuropathy, and pain. J Clin Oncol. 2012 Oct 20;30(30):3687–96.
- 353 3. Richards M, Corner J, Maher J. The National Cancer Survivorship Initiative: new and
- emerging evidence on the ongoing needs of cancer survivors. British Journal of Cancer. 2011
- 355 Nov;105(S1):S1-4.
- 356 4. Cramp F, James A, Lambert J. The effects of resistance training on quality of life in
- cancer: a systematic literature review and meta-analysis. Support Care Cancer. 2010
- 358 Nov;18(11):1367–76.
- 5. Cheema B, Gaul CA, Lane K, Fiatarone Singh MA. Progressive resistance training in
- breast cancer: a systematic review of clinical trials. Breast Cancer Res Treat. 2008 May;109(1):9–
- 361 26.
- 362 6. Spence RR, Heesch KC, Brown WJ. Exercise and cancer rehabilitation: a systematic
- 363 review. Cancer Treat Rev. 2010 Apr;36(2):185–94.
- Fuller JT, Hartland MC, Maloney LT, Davison K. Therapeutic effects of aerobic and
- resistance exercises for cancer survivors: a systematic review of meta-analyses of clinical trials. Br
- 366 J Sports Med. 2018 Oct;52(20):1311.
- Hayes SC, Spence RR, Galvão DA, Newton RU. Australian Association for Exercise
- and Sport Science position stand: optimising cancer outcomes through exercise. J Sci Med Sport.
- 369 2009 Jul;12(4):428–34.
- Rock CL, Doyle C, Demark-Wahnefried W, Meyerhardt J, Courneya KS, Schwartz
- 371 AL, et al. Nutrition and physical activity guidelines for cancer survivors. CA Cancer J Clin. 2012
- 372 Aug;62(4):243–74.
- 373 10. Salvi R, Meoli I, Cennamo A, Perrotta F, Saverio Cerqua F, Montesano R, et al.
- Preoperative high-intensity training in frail old patients undergoing pulmonary resection for

- 375 NSCLC. Open Med (Wars). 2016;11(1):443–8.
- 376 11. Edvardsen E, Skjønsberg OH, Holme I, Nordsletten L, Borchsenius F, Anderssen SA.
- High-intensity training following lung cancer surgery: a randomised controlled trial. Thorax. 2015
- 378 Mar 1;70(3):244–50.
- 379 12. Stefanelli F, Meoli I, Cobuccio R, Curcio C, Amore D, Casazza D, et al. High-
- intensity training and cardiopulmonary exercise testing in patients with chronic obstructive
- pulmonary disease and non-small-cell lung cancer undergoing lobectomy. Eur J Cardiothorac Surg.
- 382 2013 Oct;44(4):e260-265.
- Feito Y, Heinrich KM, Butcher SJ, Poston WSC. High-Intensity Functional Training
- 384 (HIFT): Definition and Research Implications for Improved Fitness. Sports (Basel). 2018 Aug
- 385 7;6(3).
- Thompson WR. WORLDWIDE SURVEY OF FITNESS TRENDS FOR 2018: The
- 387 CREP Edition. ACSM's Health & Fitness Journal. 2017 Dec;21(6):10.
- Feito Y, Hoffstetter W, Serafini P, Mangine G. Changes in body composition, bone
- metabolism, strength, and skill-specific performance resulting from 16-weeks of HIFT. PLoS ONE.
- 390 2018;13(6):e0198324.
- 391 16. Heinrich KM, Spencer V, Fehl N, Poston WSC. Mission essential fitness: comparison
- of functional circuit training to traditional Army physical training for active duty military. Mil Med.
- 393 2012 Oct;177(10):1125-30.
- 394 17. Heinrich K.M. High-intensity functional training improves functional movement and
- body composition among cancer survivors: a pilot study. 2015 Nov;
- 396 18. Bechke E, Kliszczewicz B, Feito Y, Kelemen H, Nickerson B. Resting cardiac
- 397 autonomic activity and body composition following a 16-week high-intensity functional training
- intervention in women: A pilot study. Journal of Human Sport & Exercise. 2017 Jul;12(3):680–8.
- 399 19. Ganz PA, Earle CC, Goodwin PJ. Journal of Clinical Oncology update on progress in
- 400 cancer survivorship care and research. J Clin Oncol. 2012 Oct 20;30(30):3655–6.
- 401 20. Heinrich KM., Patel PM., O'Neal JL., Heinrich BS. High-intensity compared to
- 402 moderate-intensity training for exercise initiation, enjoyment, adherence, and intentions: an
- intervention study. BMC public health. 2014;14:789.
- 404 21. Khanna N, Nesbitt L, Roghmann M-C, Tacket C. Translation of clinical research into
- practice: defining the clinician scientist. Fam Med. 2009 Jun;41(6):440–3.
- 406 22. Esculier J-F, Barton C, Whiteley R, Napier C. Involving clinicians in sports medicine

- and physiotherapy research: "design thinking" to help bridge gaps between practice and evidence.
- 408 Br J Sports Med. 2018 Oct 27;
- 409 23. Glassman G. What is CrossFit? The Crossfit Journal 2002. october 2002.
- 410 24. Claudino JG, Gabbett TJ, Bourgeois F, Souza H de S, Miranda RC, Mezêncio B, et al.
- 411 CrossFit Overview: Systematic Review and Meta-analysis. Sports Med Open. 2018 Feb 26;4(1):11.
- 412 25. What Is Fitness? [Internet]. [cited 2018 Oct 24]. Available from:
- 413 https://journal.crossfit.com/article/what-is-fitness
- Luckett T, King MT, Butow PN, Oguchi M, Rankin N, Price MA, et al. Choosing
- between the EORTC QLQ-C30 and FACT-G for measuring health-related quality of life in cancer
- clinical research: issues, evidence and recommendations. Ann Oncol. 2011 Oct;22(10):2179–90.
- 417 27. Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, et al. The
- 418 European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life
- instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar
- 420 3;85(5):365–76.
- 421 28. Fayers P. EORTC QLQ-C30 Scoring Manual The EORTC QLQ-C30. 2001:1–67.
- 422 29. Godin G, Shephard RJ. A simple method to assess exercise behavior in the
- 423 community. Can J Appl Sport Sci. 1985 Sep;10(3):141–6.
- 424 30. Jacobs DR, Ainsworth BE, Hartman TJ, Leon AS. A simultaneous evaluation of 10
- commonly used physical activity questionnaires. Med Sci Sports Exerc. 1993 Jan;25(1):81–91.
- 428 Appendices
- 429 Appendix 1

### 431 Information concerning participation in a scientific research study

- 432 Trial title:
- 433 High Intensity Functional Training in the rehabilitation of cancer survivors A pragmatic
- 434 Intervention Study 435
- We would like to ask you, if you would like to participate in a trial carried out at the Centre
- for Cancer and Health Copenhagen. The research trial is conducted by the University of
- 438 Copenhagen and physiotherapist Andreas Lund Hessner.

439

426

427

430

- Before you decide, whether you want to participate, you have to fully understand what the purpose
- of the study and why it is being conducted. Therefore, we would like to ask you to read this
- 442 participant information thoroughly.
- If you decide to participate in this study, we would like to ask you to sign a written consent
- statement. We would like to remind you that you are allowed time to consider before you decide
- whether you want to sign the written consent statement.
- Participation in this study is voluntary. At any time, and without reason you have the right to
- withdraw you consent. Withdrawing from participation in this study will not have any
- consequences for your further treatment and rehabilitation.

#### 449 Purpose

- The purpose of this study is to investigate, whether 16 weeks of High intensity functional training
- improves the health-related quality of health in cancer survivors.

452 453

454

- There is only one intervention group in this study and no control-group. There is therefore no randomization, and thus, all participants will complete 16 weeks of CrossFit-based exercise
- supervised by physiotherapists. CrossFit is a strength and conditioning program, that incorporates
- different exercise with both free weights and bodyweight movements.

457 458

#### Plan for study period

- With your consent you agree to participate in 16-week weeks of group-based exercise including two
- 460 weekly exercise sessions.
- Prior to starting the intervention, we are going to ask you to complete a questionnaire with
- questions concerning cancer treatment, symptoms and physical activity level.
- 463 Immediately following 16-week intervention period you will receive another questionnaire. Three
- and 12 months following completion of the intervention period we will ask you to complete two
- 465 identical questionnaires.
- 466 Following completion, the results of this trial will be published in scientific journals and will be
- presented at national medical conferences. All your personal information in this study is
- anonymised.

469 470 471

472

473

474

475

#### Your health information

All outcome in this study is going to be collected through questionnaires. This means that we will only collect information about you through these electronic questionnaires. Thus, there will not be collected information about you or your health from medical records of any kind.

476

477 478

479

480

- If you consent to participate in this study, we will ask you for your e-mail address and as previously stated you will be asked to complete a total of four questionnaires. If you consent to participate we
- will in within the next two days send you the baseline questionnaire electronically.
- We ask you to complete this questionnaire before your first High intensity functional training session in the intervention.

484 485

#### Relevance and benefits of the study

- 486 You will contribute to new knowledge and insights concerning the physical rehabilitation of people
- living with cancer, including the types of exercise, that might be beneficial for cancer survivors.

488 489

Potential side-effects, risks and complications

| | Non serious potential side-effects | Serious | Long term risks |
|---|---|---|---|
| Side-effects | Muscle and joint pain | None | None |
| | Potential passing discomfort during the | | |
| | exercise sessions such as shortness of breath | | |
| | or dizzyness | | |

490 491

492

There may occur risks associated with this study, that we do not yet know about. We ask you to notify us, if you are to experience any health problems or concerns, during your participation in the study.

493 494 495

496 497

498

#### **Exclusion or interruption of study**

If the health personnel at Centre for Cancer and Health Copenhagen assess that there may be health circumstances, which may imply that your continuation in this study may be associated with any type of risk, your participation in this study will be terminated. In this case the health personal will assist you in finding the best course of action.

499 500 501

#### Information about economic/financial conditions

No financial benefits are associated with your participation in this study.

502503504

505

#### Access to study results

- One peer reviewed article will be published in a scientific journal, during the fall of 2020.
- The results of this study will upon publication be communicated to various media and through the website of Centre for Cancer and health Copenhagen.
- We hope that you through this information have received adequate insights into what it entails to
- participate in this study, and that you feel appropriately informed to make the decision whether to
- participate. We ask you to read the attached amendment concerning "subjects rights in health
- scientific research projects".
- If you would like more information about the study, we recommend you to contact project leader

513

- 514 Andreas Lund Hessner
- 515 E-Mail: <u>hessnerfysioterapi@gmail.com</u>
- 516 Telephone: 51964161

Best regards,

517

Andreas Lund Hessner, PT, MSc.

519520

- 521522
- 523
- 524